CLINICAL TRIAL: NCT07343362
Title: Zeus Sleep Technology: A UK-based Multi-centre Randomised Controlled Trial Using Transcutaneous Electrical Stimulation in Patients With Obstructive Sleep Apnoea (TESLA)
Brief Title: Transcutaneous Electrical Stimulation in Patients With Obstructive Sleep Apnoea
Acronym: TESLA-MICRON
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeus Sleep Ltd (Industry)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); King's College London (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Queen Victoria Hospital NHS Foundation Trust (Other Government); The Queen Elizabeth Hospital (Other); Imperial College Healthcare NHS Trust (Other); AintreeNHSTrust (Unknown); University of Southampton (Other); Royal Papworth Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZEUSi4i-1.0-03/12/25; NIHR209411 (Other Grant/Funding Number: National Institute for Health and Care Research (NIHR))
Record Dates: First submitted 2025-12-17; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: CPAP; Continuous Positive Airway Pressure; Hypoglossal Nerve Stimulation; non-CPAP therapy; sleep-disordered breathing; TESLA-MICRON; Zeus Sleep Technology; transcutaneous electrical stimulation; Zeus Sleep Ltd
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Two-group, parallel, interventional randomized controlled trial
  Sample Size Calculation The sample size estimates were based on the previous trial by Ratneswaran et al. 2023 (eClinMed) where the primary outcome was change in mean apnea-hypopnea index (AHI) at 3-months between two trial arms. The difference adjusted for the baseline value was -7.0 (95% CI: -15.7;1.8), and the common standard deviation within group was 18. Using these estimates for an analysis of covariance, sample sizes of 74, and 74 are required from each of the 2 trial groups whose means are to be compared. The covariate was assumed to have an R-squared of 0.30. The total sample of 148 subjects achieves 80% power to detect the differences described by Ratneswaran between the two means, with 0.05 00 significance level. Allowing for 20% dropout the sample required is 186 participants in the two groups.
Masking Description: The analysis of the sleep studies will be undertaken by an independent party (outsourced data provider) and allocation to the RCT arms will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Continuous Positive Airway Pressure (CPAP)
  Interventions: Device: CPAP
- Intervention (Experimental): Transcutaneous Electrical Stimulation (ZeusOSA)
  Interventions: Device: ZeusOSA

INTERVENTIONS:
Device: ZeusOSA — Transcutaneous electrical stimulation in sleep apnoea (TESLA) in the submittal area, provided by the ZeusSleep device when asleep.
  Arms: Intervention
Device: CPAP — Continous positive airway pressure (CPAP) when asleep
  Arms: Usual Care

SUMMARY:
The objective of this trial is to assess efficacy and compliance of transcutaneous electrical stimulation of the upper airway dilator muscles in patients with obstructive sleep apnoea (TESLA) who do not tolerate continuous positive airway pressure (CPAP) therapy over a period of 3-months in the community and compare results against usual care (ongoing CPAP therapy), evaluate acceptability, comfort and adverse events, and record outcomes for provision of the health economics analysis. The proposed study will provide us with data about the efficacy of the domiciliary use of the intervention from a UK-based prospective, multi-centre and randomised controlled trial (Phase III). We will understand whether the primary outcome parameter, the apnoea hypopnea index (AHI), or the secondary outcomes (e.g., 4% oxygen desaturation index (ODI), the Epworth Sleepiness Scale (ESS), compliance and comfort, functional outcome of sleep questionnaires (FOSQ), European Quality of Life Questionnaire (EQ-5D)) are suitable measures to assess control of OSA using TESLA within reasonable acceptance for the patients to provide the analysis of healthcare resource usage for assessment of cost-efficacy and quality-adjusted life years (QALYs). Responder analysis will provide insights into gender, socio-economic background and endotypes to predict who most suitably benefits from this treatment.

DETAILED DESCRIPTION:
The TESLA-MICRON study is a UK-based, prospective, multi-centre, randomised controlled trial designed to evaluate the use of an investigational medical device, ZeusOSA, for the treatment of obstructive sleep apnoea in adults with poor adherence to continuous positive airway pressure (CPAP) therapy.

ZeusOSA uses gentle stimulation through the skin similar to that of a TENS machine. The device features a U-shaped lightweight silicone pad with a disposable adhesive hydrogel electrode pad (single-use) that delivers mild transcutaneous electrical nerve stimulation (TENS) to activate the hypoglossal nerve, thereby stimulating muscles to contract, particularly those associated with opening the airways (e.g., genioglossus muscle). Application of regular electrical pulses to these muscles help to maintain an open airway. The upper airway muscles might otherwise relax with sleep onset and cause vibrations and collapse in the throat whilst breathing, manifesting as snoring or sleep apnoea's or hypopneas. The stimulation level is customisable from level 1 (milder stimulation) to level 10 (stronger stimulation).

186 participants will be recruited with a prior diagnosis of obstructive sleep apnoea and low CPAP adherence at follow up (less than 4 hours/night) will be randomly assigned in a 1:1 ratio to either the intervention group or a usual care group. Recruitment will focus on a balanced ratio of men and women, as women are typically under-represented in studies of OSA and, due to a slim neck / collar size in comparison to men, likely to be responders to the TESLA treatment. Participants allocated to the intervention group will use the investigational medical device, ZeusOSA, which delivers transcutaneous electrical stimulation to the upper airway dilator muscles during sleep. The device is intended for nightly use at home over a three-month period. Participants in the usual care group will continue with ongoing CPAP therapy in accordance with current clinical practice.

All participants will undergo baseline assessments prior to randomisation, including a home-based sleep study conducted without treatment. Follow-up will include a scheduled telephone contact at approximately six weeks and a repeat assessment at three months, including a further home-based sleep study conducted with the assigned treatment and receive standard advice on sleep hygiene and lifestyle measures. The patients will then be referred for follow up to standard care in the outpatient setting at their respective sleep centre. The trial duration including recruitment is 3 years.

The study will assess the therapeutic effects of the investigational medical device on sleep-related outcomes and symptoms, as well as participant-reported quality of life. Additional objectives include evaluation of treatment adherence, comfort and acceptability of use, and monitoring of adverse events. Data collected during the study will also be used to support an assessment of healthcare resource use associated with the intervention.

The study is designed to reflect real-world use of the investigational medical device in a domiciliary setting and to identify patient characteristics associated with response to treatment. Results from this trial will inform the future clinical and regulatory development of the device for the management of obstructive sleep apnoea.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants (≥18 years) who have OSA with an AHI between 5-40 events/hour.
2. If participant fails to use CPAP sufficiently with less than 4 hours/night.
3. Adults with a body mass index (BMI) of 18.5-32.0 kg/m2,
4. Adults without significant anatomical obstruction in the upper airway (e.g., normal sized tonsils).
5. Able to provide informed consent.

Exclusion Criteria:

1. Adults with no OSA (AHI <5/h), or with very severe OSA (AHI>40/hour).
2. Adults who are cachectic (BMI <18.5 kg/m2) or very obese (BMI >32 kg/m2).
3. Hypercapnic patients (pCO2>6.0 kPa) or those with other features of obesity hypoventilation syndrome (elevated bicarbonate, HCO3- >28mmol/L).
4. Adults should not have significantly enlarged tonsils (size 3-4)
5. Adults with polyps or adenoids, hypoglossal nerve palsy,
6. Adults with notable medical co-morbidities that could potentially impact participation in or the achievement of the study's objectives (e.g., significant heart failure (New York Heart Association, NYHA class III-IV), recent myocardial infarction (within 3 months) and significant cardiac arrhythmias, uncontrolled hypertension).
7. Participants with active psychiatric disease.
8. Adults with significant metal implants in head / neck, or cardiac/other pacemakers.
9. Participants who are physically incapacitated such as to manoeuvre the Zeus device
10. Adults who do not have access to a smartphone and/or internet data at home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2026-07-16 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea-index (AHI) | Baseline to 3 months
  Number of respiratory events per hour measured by home-based sleep study.

SECONDARY OUTCOMES:
Epworth Sleepiness Scale (ESS) | Baseline to 3 months
  Daytime sleepiness measured using the Epworth Sleepiness Scale (score range 0-24, with higher scores indicating greater sleepiness).
EQ-5D Index Score | Baseline to 3 months
  Health-related quality of life measured using the EQ-5D descriptive system (index score 0-1).
EQ-5D Visual Analogue Scale (VAS) Score | Baseline to 3 months
  Self-rated health measured using the EQ-5D visual analogue scale (0-100, with higher scores indicating better perceived health).
Functional Outcome of Sleep Questionnaire (FOSQ-10) Score | Baseline to 3 months
  Sleep-related functional status measured using the FOSQ-10, with higher scores indicating better functional outcomes.
Snoring Duration | Baseline to 3 months
  Total duration of snoring measured during sleep, expressed in minutes.
Snoring Intensity | Baseline to 3 months
  Average snoring intensity measured in decibels during sleep.
Adherence Average hours/night | Baseline to 3 months
  Average nightly usage (hours) of the assigned treatment.
Adherence - Percentage of Nights Used | Baseline to 3 months
  Percentage of nights the assigned treatment was used during the study period.

OTHER OUTCOMES:
SHER15 criteria defining responders to treatment | 3-months
  Reduction of AHI of more than 50% to below 15 events per hour, or normal (below 5 per hour);
SHER20 criteria defining responders to treatment | 3-months
  Reduction of AHI of more than 50% to below 20 events per hour, or normal (below 5 per hour);
Gender-related response | 3-months
  Responder rate according to gender (male vs female responders, percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Steier, PhD, Study Chair — Guy's & St Thomas' NHS Foundation Trust, London, UK

IPD SHARING:
Plan to Share IPD: Undecided
Pending ethics approval and medio-legal framework (GDPR)